CLINICAL TRIAL: NCT05428085
Title: The Relationship Between the Digital Media Usage With Impulsivity and Attention Deficit in Children With Early Intervention
Brief Title: Digital Media Usage With Impulsivity and Attention Deficit in Children
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Hsinchieh Lee, Taipei Medical University Shuang Ho Hospital, Taipei Medical University Shuang Ho Hospital
Other Study IDs: N202204077
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Attention-Deficit-Disordered Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers whose children are currently receiving early treatment: Individual caregivers were interviewed through paper questionnaires to assess children's and families' digital media usage habits, children's activity levels, and parental stress. Pearson's Chi-Square test and liner regression was used for analysis.

SUMMARY:
To explore the relationship between children's digital media usage and attention, activity, parenting pressure; to explore the relationship between family basic data factors and screen usage.

DETAILED DESCRIPTION:
Background: Digital products are inseparable from life. Parents may feel that teaching materials are educational because of their high availability.Meaning, busy work, helping to share care or short respite, etc., and providing digital products for children, it is very important to understand children's behavior, usage habits, and the relationship between parents.According to the American Academy of Pediatrics, parents should limit their exposure to most types of screen time until the child is 2 years old , and children 2-5 years old should be less than one hour per day, and it is recommended to watch high Quality program content, accompanied by adults. The standards for screen time in various countries generally follow this policy.However, many studies have found that most children spend far more screen time than recommended guidelines. Research in Canada and the United States indicates that children aged three to five spend more than two hours a day on average. According to a tracking study, children aged three to five were surveyed on their In terms of screen use, it was found that compared with children who watched less than half an hour, children who used more than two hours a day had more significant implicit and explicit behavioral problems, namely withdrawal, nervousness, anxiety, irritability and attention deficit, and restless behavior.

Objective: To explore the relationship between children's digital media usage and attention, activity, parenting pressure; to explore the relationship between family basic data factors and screen usage.

Methods: Individual caregivers were interviewed through paper or electronic questionnaires to assess children's and families' digital media usage habits, children's activity levels, and parental stress. The following assessment tools were used. Including digital media use survey at home (refer to Surveillance of digital-Media habits in earLy childhood Questionnaire, SMALLQ™), Chinese version of parental child activity scale (Werry-Weiss Peters Activity Scale Chinese version, WWPAS), parental stress scale brief Form (Parenting Stress Index: Short form, PSI/SF)

ELIGIBILITY:
Inclusion Criteria:

* Caregivers whose children are currently receiving early treatment and who can cooperate with the questionnaire;
* The child's family has the habit of using digital media devices;
* The child's main complaints include inattention and impulsivity;
* The child's age is 3 to 6 years old.

Exclusion Criteria:

* The child has other specific diagnosed diseases, such as autism group, sensory disorder, known genetic and genetic diseases, etc.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Children who spent screen time more than two hours a day had more significant implicit and explicit behavioral problems, namely withdrawal, nervousness, anxiety, irritability and attention deficit, and restless behavior.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Surveillance of digital-Media habits in earLy childhood Questionnaire, SMALLQ™ | Baseline at first evaluate time
  An survey used to estimate the weekday & weekend parent-reported on-screen & off-screen media habits of preschoolers, among other things. The information including three segments: (i) digital media use, parent concern, knowledge and practice of guidelines, outside of school on weekday and weekend; (ii) non-digital media habits: indoor and outdoor play, day time naps, non-screen reading, and drawing; (iii) parent educational attainment and household income, additional child information: height, weight, wearing spectacles or not, and night-time sleep.

SECONDARY OUTCOMES:
Werry-Weiss Peters Activity Scale Chinese version, WWPAS | Baseline at first evaluate time
  It is a 27 items inventory completed by parents, aimed at evaluating the child's activity level in a family context, in various situations of daily life (e.g., during meals, watching television, while playing, in activities abroad). The total result is obtained by adding directly the scores of all the items and represents a general measure of the child's activity level. Parents rated the frequency of their child's behaviors as occurring "none," "some," or "much of the time" . However, interparent interrater reliability was reported to be good (Barkley, 1988). No information regarding the test-retest reliability or internal consistency was located (Barkley, 1988).
Parental stress scale brief Form | Baseline at first evaluate time
  The scale assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. emotional benefits, personal development) and negative aspects of parenthood (e.g. demands on resources, feelings of stress). It contains various measures of stress, emotion and role satisfaction, including perceived stress, work/family stress, loneliness, anxiety, guilt, marital satisfaction/commitment, job satisfaction, and social support. The PSI has 36 items with a 5-point Likert scale, with response options ranging from "strongly agree" to "strongly disagree." Responses on the measure are summed to create a total stress (TS) composite, which provides an indication of the amount of stress adults are experiencing due to their role as a parent (Abidin 1995). Internal consistency reliability was high for TS (α = .90).

CONTACTS AND LOCATIONS:
Overall Officials: Hsinchieh Lee, master, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chia, M., Tay, L. Y., & Chua, T. B. K. (2019). The development of an online surveillance of digital media use in early childhood questionnaire-SMALLQ™-for Singapore.
- [Background] Huang Y, Yan Q, Tong L. Reliability and validity of an observation-based parent-child interaction rating scale for Chinese children aged 0-6 years. Psychol Assess. 2022 May;34(5):e45-e54. doi: 10.1037/pas0001121. Epub 2022 Mar 24. PMID 35324253
- [Background] Werry-Weiss-Peters Activity Scale, W. W. P. Center for Research in Neuropsychology and Cognitive Behavioral Intervention.
- [Background] Abidin, R. R. (1995). Parenting Stress Index (PSI) manual . Odessa, FL: Psychological Assessment Resources.
- [Background] Tamana SK, Ezeugwu V, Chikuma J, Lefebvre DL, Azad MB, Moraes TJ, Subbarao P, Becker AB, Turvey SE, Sears MR, Dick BD, Carson V, Rasmussen C; CHILD study Investigators; Pei J, Mandhane PJ. Screen-time is associated with inattention problems in preschoolers: Results from the CHILD birth cohort study. PLoS One. 2019 Apr 17;14(4):e0213995. doi: 10.1371/journal.pone.0213995. eCollection 2019. PMID 30995220
- [Background] Poitras VJ, Gray CE, Janssen X, Aubert S, Carson V, Faulkner G, Goldfield GS, Reilly JJ, Sampson M, Tremblay MS. Systematic review of the relationships between sedentary behaviour and health indicators in the early years (0-4 years). BMC Public Health. 2017 Nov 20;17(Suppl 5):868. doi: 10.1186/s12889-017-4849-8. PMID 29219092
- [Background] Beal JA. Screen Time and Toddlers: New Evidence on Potentially Negative Effects. MCN Am J Matern Child Nurs. 2020 Jul/Aug;45(4):241. doi: 10.1097/NMC.0000000000000632. No abstract available. PMID 32604184
- [Background] Radesky JS, Christakis DA. Increased Screen Time: Implications for Early Childhood Development and Behavior. Pediatr Clin North Am. 2016 Oct;63(5):827-39. doi: 10.1016/j.pcl.2016.06.006. PMID 27565361
- [Background] Madigan S, Browne D, Racine N, Mori C, Tough S. Association Between Screen Time and Children's Performance on a Developmental Screening Test. JAMA Pediatr. 2019 Mar 1;173(3):244-250. doi: 10.1001/jamapediatrics.2018.5056. PMID 30688984
- [Background] Kids & Tech: Tips for Parents in the Digital Age. HealthyChildren.org. (n.d.). https://www.healthychildren.org/English/family-life/Media/Pages/Tips-for-Parents-Digital-Age.aspx.
- [Background] American Academy of Pediatrics Healthy Children. Org. (2016). How to develop a family media plan [Website]. https://www.healthychildren.org/English/family-life/Media/Pages/How-to-Make-a-Family-Media-Use-Plan.aspx
- [Background] Australian Government Department of Health and Ageing (DoHA) (2011). Get Up and Grow: Healthy Eating and Physical Activity for Early Childhood-Family Book. Retrieved 20 February 2022, from www.health.gov.au/internet/publications/publishing.nsf/Content/gug-family-toc.
- [Background] Xie G, Deng Q, Cao J, Chang Q. Digital screen time and its effect on preschoolers' behavior in China: results from a cross-sectional study. Ital J Pediatr. 2020 Jan 23;46(1):9. doi: 10.1186/s13052-020-0776-x. PMID 31973770
- [Background] Reid Chassiakos YL, Radesky J, Christakis D, Moreno MA, Cross C; COUNCIL ON COMMUNICATIONS AND MEDIA. Children and Adolescents and Digital Media. Pediatrics. 2016 Nov;138(5):e20162593. doi: 10.1542/peds.2016-2593. PMID 27940795
- [Background] Vandewater EA, Rideout VJ, Wartella EA, Huang X, Lee JH, Shim MS. Digital childhood: electronic media and technology use among infants, toddlers, and preschoolers. Pediatrics. 2007 May;119(5):e1006-15. doi: 10.1542/peds.2006-1804. PMID 17473074
- [Background] Rideout, V. (2011). Zero to eight: Children's media use in America. Common Sense Media.